CLINICAL TRIAL: NCT06925776
Title: Community Health Workers in an Interdisciplinary Outpatient CKD Clinic to Optimize Social Care Navigation, Patient Engagement, and Home Dialysis Utilization- the CHOOSE Home Trial
Brief Title: Community Health Workers in an Interdisciplinary Outpatient CKD Clinic to Optimize Social Care Navigation, Patient Engagement, and Home Dialysis Utilization
Acronym: CHOOSE Home
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2025-16868; 1R01DK140574-01 (NIH)
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Kidney Replacement Therapy
Keywords: Community Health Worker; Interdisciplinary Care; Kidney Replacement Therapy; home dialysis; Health-Related Social Needs; patent engagement; Hemodialysis; home hemodialysis; peritoneal dialysis
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Pilot, pragmatic, randomized, parallel two-arm single site trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHW facilitated social care navigation and peer support as part of IDC (Other): Patients will receive community health worker (CHW) facilitated social care navigation and peer support around kidney replacement therapy (KRT) decision-making as part of their interdisciplinary care (IDC) for CKD, up to 1 year.
  Participants will complete surveys, questionnaires, or interviews at baseline, 6 months, and 12 months.
  Interventions: Other: CHOOSE Home Intervention
- IDC alone (Other): Patients will receive IDC (Interdisciplinary Care) only. They will not receive CHW (Community Health Worker) facilitated peer support and social care navigation.
  Participants will complete surveys, questionnaires, or interviews at baseline, 6 months, and 12 months.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: CHOOSE Home Intervention — Integration of a CHW (Community Health Worker) in the CKD (Chronic Kidney Disease) care process to augment patient engagement and address HRSNs (Health-Related Social Needs) within the context of an IDC (Interdisciplinary Care) CKD clinic. The multifaceted components of the intervention are tailored to address key care delivery and social barriers to home dialysis utilization before implementation.
  Other Names: CHW Intervention; CHW + IDC Intervention; IDC + CHW
  Arms: CHW facilitated social care navigation and peer support as part of IDC
Other: Usual Care — This is the usual interdisciplinary care that patients would typically receive for their chronic kidney disease. A key missing factor here is the lack of a community health worker. Patients in this group will be screened for health-related social needs and receive general information on ways to access social services from a study coordinator. Patients will not receive facilitated peer support and social care navigation from the Community Health Worker.
  Other Names: Control Group
  Arms: IDC alone

SUMMARY:
The goal of this clinical trial is to learn if this intervention (the CHOOSE Home intervention) is feasible and may lead to more home dialysis usage in a high-risk patient population. The main questions it aims to answer are:

* Will there be an increase in home dialysis selection or initiation over study follow up?
* Will there be a change in patient reported status of Health-Related Social Needs (HRSNs) and patient engagement at 1 year follow up?

Researchers will compare the intervention group that will include interdisciplinary care (IDC) and the integration of a Community Health Worker (CHW) into the chronic kidney disease (CKD) care process to the IDC only control group. The research team will assess whether the intervention led to better social care navigation, enhanced patient engagement, and increased home dialysis use.

DETAILED DESCRIPTION:
The overarching aims of the study are to 1) utilize a community- engaged approach with input from diverse community partners to refine the CHOOSE Home Trial; and 2) evaluate the feasibility, acceptability, and possible effect of the CHOOSE Home Intervention. Feasibility and acceptability will be evaluated using complementary quantitative and qualitative measures and organized into the dimensions of the RE-AIM framework. The investigator team hypothesizes that the CHOOSE Home intervention may lead to increased home dialysis utilization by more effectively addressing health-related social needs and fostering greater patient engagement. This proposal brings together experts in CKD care, SDOH, health equity, implementation and community-engaged research. The results will be used to inform further studies in CKD care delivery to reduce health inequities in home dialysis use and improve the quality of life for patients with CKD.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Advanced CKD (defined by estimated glomerular filtration rate (eGFR) of 25 ml/min/1.73m2 or less using the 2021 Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation)
* English or Spanish speaking
* Provide informed consent
* Followed by a nephrologist at Montefiore and seen within last 12 months
* Willing to receive interdisciplinary care (i.e., nurse practitioner facilitated CKD education and care coordination)

Exclusion Criteria:

* Active malignancy
* Anticipated survival is less than 1 year as determined by the patient's treating nephrologist
* Opting to do medical management only (non- dialysis supportive care) for management of their kidney failure
* Plan to relocate outside of New York City within the next 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-12-12 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Selection or Initiation of Home Dialysis | 1 year study follow up period
  The percentage of patients who select or initiate home dialysis in each study arm will be summarized by study arm. To account for patients who may not progress to end-stage kidney disease (ESKD) within one year, this percentage will be defined as the sum of non-ESKD patients choosing home dialysis and ESKD patients who start home dialysis, divided by the total patients in each group.

SECONDARY OUTCOMES:
Change in Patient Activation Measure Scores | From baseline to 6 months and baseline to 1 year
  Change in Patient Activation Measure (Patient Engagement) will be assessed by assessment of the Patient Activation Measure (PAM) survey at baseline, 6 months, and 1 year.
  The PAM is a 13-item survey designed to assess a patient's knowledge, beliefs, confidence, and skills about managing one's healthcare. Each item is scored on a 4-point Likert scale ranging from 1 ("Strongly disagree") to 4 ("Strongly Agree"). Raw scores are transformed to a scale with a theoretical range of 0-100, based on calibration tables, with higher PAM scores indicating higher levels of patient activation.
  For purposes of this study, change from baseline to 6 months and 1 year will be assessed, and positive percentage scores will indicate increased patient activation.
  The percentage of patients in each arm with a 6-point PAM increase over a period of 6-12 months will be summarized by study arm.
Change in patient-reported status of Health-related social needs (HRSNs) | From baseline to 6 months and baseline to 1 year
  HRSNs will be assessed by the by administration of the Accountable Health Communities Health-Related Social Needs (AHC-HRSN) survey at baseline and 1 year.
  The AHC-HRSN is a 26-item screening tool designed to help providers identify patients' needs. This study will focus on five core domains captured in the first 10-items of the screening tool. The five core domains are housing instability, food insecurity, transportation problems, interpersonal safety, and utility help. If a patient answers positively to any domain(s) and desires assistance, they are considered to have that corresponding health-related social need.
  Change in HRSN status (i.e., resolved/progress made or no progress) from baseline to 6 months and 1 year will be categorized and summarized by study arm.

CONTACTS AND LOCATIONS:
Overall Officials: Tanya S Johns, MD, MHS, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with NIH guidelines, the study team will share data with qualified investigators whose research protocols have been approved by their institutions' Institutional Review Boards. The final dataset will include qualitative and quantitative data including anonymized transcripts, socio-demographics, medical history, social history, and clinical outcomes data. The dataset will be stripped of all personal identifiers according to HIPAA and the Common Rule. The investigator team plans to submit anonymized data to a generalist repository, Vivli, that is participating in the NIH Generalist Repository Ecosystem Initiative (GREI) so that it can be made available to other investigators under an NIH-approved data-sharing agreement that ensures that: (1) data is used only for research purposes and does not identify individual participants; (2) data is handled in a secure and confidential way; and (3) data is destroyed or returned after analyses are completed.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Following publication, time frame to be determined
Access Criteria: Data will be shared with qualified research investigators whose research protocols have been approved by their institutions' Institutional Review Boards.
URL: https://vivli.org

REFERENCES:
- [Background] United States Renal Data System. 2022 USRDS Annual Data Report: Epidemiology of kidney disease in the United States. National Institutes of Health, National Institute of Diabetes and Digestive and Kidney Diseases, Bethesda, MD, 2022.
- [Background] Francois K, Bargman JM. Evaluating the benefits of home-based peritoneal dialysis. Int J Nephrol Renovasc Dis. 2014 Dec 4;7:447-55. doi: 10.2147/IJNRD.S50527. eCollection 2014. PMID 25506238
- [Background] Johns TS, Prudhvi K, Motechin RA, Sedaliu K, Estrella MM, Stark A, Bauer C, Golestaneh L, Boulware LE, Melamed ML. Interdisciplinary Care and Preparedness for Kidney Failure Management in a High-Risk Population. Kidney Med. 2022 Mar 17;4(5):100450. doi: 10.1016/j.xkme.2022.100450. eCollection 2022 May. PMID 35479194
- [Background] Johns TS, Yee J, Smith-Jules T, Campbell RC, Bauer C. Interdisciplinary care clinics in chronic kidney disease. BMC Nephrol. 2015 Oct 12;16:161. doi: 10.1186/s12882-015-0158-6. PMID 26458811
- [Background] Cho EJ, Park HC, Yoon HB, Ju KD, Kim H, Oh YK, Yang J, Hwang YH, Ahn C, Oh KH. Effect of multidisciplinary pre-dialysis education in advanced chronic kidney disease: Propensity score matched cohort analysis. Nephrology (Carlton). 2012 Jul;17(5):472-9. doi: 10.1111/j.1440-1797.2012.01598.x. PMID 22435951
- [Background] Hsu HT, Chiang YC, Lai YH, Lin LY, Hsieh HF, Chen JL. Effectiveness of Multidisciplinary Care for Chronic Kidney Disease: A Systematic Review. Worldviews Evid Based Nurs. 2021 Feb;18(1):33-41. doi: 10.1111/wvn.12483. Epub 2020 Nov 28. PMID 33247619
- [Background] Peeters MJ, van Zuilen AD, van den Brand JA, Bots ML, van Buren M, Ten Dam MA, Kaasjager KA, Ligtenberg G, Sijpkens YW, Sluiter HE, van de Ven PJ, Vervoort G, Vleming LJ, Blankestijn PJ, Wetzels JF. Nurse practitioner care improves renal outcome in patients with CKD. J Am Soc Nephrol. 2014 Feb;25(2):390-8. doi: 10.1681/ASN.2012121222. Epub 2013 Oct 24. PMID 24158983
- [Background] Manns BJ, Garg AX, Sood MM, Ferguson T, Kim SJ, Naimark D, Nesrallah GE, Soroka SD, Beaulieu M, Dixon SN, Alam A, Allu S, Tangri N. Multifaceted Intervention to Increase the Use of Home Dialysis: A Cluster Randomized Controlled Trial. Clin J Am Soc Nephrol. 2022 Apr;17(4):535-545. doi: 10.2215/CJN.13191021. Epub 2022 Mar 21. PMID 35314481
- [Background] Molnar AO, Harvey A, Walsh M, Jain AK, Bosch E, Brimble KS. The WISHED Randomized Controlled Trial: Impact of an Interactive Health Communication Application on Home Dialysis Use in People With Chronic Kidney Disease. Can J Kidney Health Dis. 2021 Jun 4;8:20543581211019631. doi: 10.1177/20543581211019631. eCollection 2021. PMID 34158965
- [Background] Sanders KA, Whited A, Martino S. Motivational interviewing for patients with chronic kidney disease. Semin Dial. 2013 Mar-Apr;26(2):175-9. doi: 10.1111/sdi.12052. Epub 2013 Feb 14. PMID 23406198
- [Background] Lunardi LE, Hill K, Xu Q, Le Leu R, Bennett PN. The effectiveness of patient activation interventions in adults with chronic kidney disease: A systematic review and meta-analysis. Worldviews Evid Based Nurs. 2023 Jun;20(3):238-258. doi: 10.1111/wvn.12634. Epub 2023 Mar 12. PMID 36906914
- [Background] Fiori KP, Rehm CD, Sanderson D, Braganza S, Parsons A, Chodon T, Whiskey R, Bernard P, Rinke ML. Integrating Social Needs Screening and Community Health Workers in Primary Care: The Community Linkage to Care Program. Clin Pediatr (Phila). 2020 Jun;59(6):547-556. doi: 10.1177/0009922820908589. Epub 2020 Mar 5. PMID 32131620
- [Background] Creswell JW. Qualitative inquiry and research design: Choosing among five approaches, 2nd ed. Thousand Oaks, CA, US: Sage Publications, Inc, 2007.
- [Background] Bronfenbrenner U. Toward an experimental ecology of human development. Am Psychol. 1977;32:513-531. doi:10.1037/0003-066X.32.7.513
- [Background] Weinstein ND. The precaution adoption process. Health Psychol. 1988;7(4):355-86. doi: 10.1037//0278-6133.7.4.355. PMID 3049068
- [Background] Weinstein ND, Sandman PM. A model of the precaution adoption process: evidence from home radon testing. Health Psychol. 1992;11(3):170-80. doi: 10.1037//0278-6133.11.3.170. PMID 1618171
- [Background] Glasgow RE, Harden SM, Gaglio B, Rabin B, Smith ML, Porter GC, Ory MG, Estabrooks PA. RE-AIM Planning and Evaluation Framework: Adapting to New Science and Practice With a 20-Year Review. Front Public Health. 2019 Mar 29;7:64. doi: 10.3389/fpubh.2019.00064. eCollection 2019. PMID 30984733